CLINICAL TRIAL: NCT02427243
Title: A Phase 1, Single-Dose, Randomized, Open-Label, Parallel Group Study to Assess the Relative Bioavailability and Tolerability of Two Formulations of Crenezumab in Healthy Subjects Following Subcutaneous Administration
Brief Title: A Study in Healthy Volunteers to Assess the Relative Bioavailability and Tolerability of Two Crenezumab Formulations Following Administration of a Single Subcutaneous Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP29172
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — crenezumab; rhoA GTP-Binding Protein

ARMS (2):
- Crenezumab Formulation 2 (Experimental): A single dose given as two subcutaneous injections on Day 1
  Interventions: Drug: Crenezumab
- Crenezumab Formulation 3 (Experimental): A single dose given as two subcutaneous injections on Day 1
  Interventions: Drug: Crenezumab

INTERVENTIONS:
Drug: Crenezumab
  Other Names: RO5490245 or MABT5102A (formerly)
  Arms: Crenezumab Formulation 3
Drug: Crenezumab
  Other Names: RO5490245 or MABT5102A (formerly)
  Arms: Crenezumab Formulation 2

SUMMARY:
To assess the relative bioavailability and tolerability of two different formulations of crenezumab in approximately 60 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 18 to 65 years of age at Screening, inclusive
* Body mass index (BMI) 18.5 to 32 kg/m^2, inclusive
* Body weight 50 to 100 kg, inclusive
* Females must be of non-childbearing potential
* Males of reproductive potential must agree to remain abstinent or must be using highly effective contraception and must avoid sperm donation, from Screening until at least 8 weeks after the last study drug administration or until study completion, whichever is later

Exclusion Criteria:

* Significant medical history, psychiatric disorder, or acute infection at Screening (as determined by Investigator)
* History of alcoholism or drug addiction within 6 months prior to CRU Check-in
* Use of tobacco or nicotine-containing products from 6 months prior to CRU Check-in and during the study
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred wtihin 30 days or 5 half-lives, whichever is longer, prior to CRU Check-in

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of crenezumab (Cmax, tmax, AUC0-last, AUC(0-infinity), Vz/F, CL/F, Apparent terminal elimination rate constant, and t1/2) | Day 1 through Day 85 or early termination

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events | Consent through Day 85 or early termination
Incidence of anti-therapeutic antibodies (ATAs) to crenezumab | From Day 1 (Predose) through Day 85 or early termination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Evansville, Indiana
  - Dallas, Texas